CLINICAL TRIAL: NCT01900717
Title: Evaluation of Bevacizumab in Combination With First-Line Chemotherapy in Patients Aged 75 Years of Older With Metastatic Colorectal Adenocarcinoma
Brief Title: Evaluation of Bevacizumab in Combination With First-Line Chemotherapy in Patients Aged 75 Years of Older With Metastatic Colorectal Adenocarcinoma (Prodige20)
Acronym: Prodige20
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Bedenne PHRC K 2010.; 2010-022080-34 (EudraCT Number)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Colorectal Adenocarcinoma
MeSH Terms: interventions — Bevacizumab

ARMS (2):
- chimiotherapy alone (Active Comparator): * LV5FU2 simplified,
  * 5-fluorouracil/leucovorin with oxaliplatin 4 (FOLFOX) simplified,
  * fluorouracil, leucovorin, and irinotecan(FOLFIRI) modified.
  Interventions: Drug: LV5FU2 simplified, FOLFOX 4 simplified, FOLFIRI modified
- chemiotherapy + bevacizumab 5 mg/kg/ 2 weeks (Experimental): * LV5FU2 simplified,
  * FOLFOX 4 simplified,
  * FOLFIRI modified.
  * Bevacizumab 5 mg/kg/ 2 weeks
  Interventions: Drug: LV5FU2 simplified,FOLFOX 4 simplified, FOLFIRI modified, Bevacizumab 5 mg/kg/ 2 weeks

INTERVENTIONS:
Drug: LV5FU2 simplified, FOLFOX 4 simplified, FOLFIRI modified
  Arms: chimiotherapy alone
Drug: LV5FU2 simplified,FOLFOX 4 simplified, FOLFIRI modified, Bevacizumab 5 mg/kg/ 2 weeks
  Arms: chemiotherapy + bevacizumab 5 mg/kg/ 2 weeks

SUMMARY:
To evaluate tolerance to and efficacy of bevacizumab in the treatment of MCRC in elderly patients, we propose a phase II randomised study comparing a chemotherapy + bevacizumab arm with a chemotherapy alone arm in the first-line treatment of MCRC in patients aged 75 years and older.

This study is destined to continue as a phase III trial if both arms meet the selection criteria to show or not the benefits of treatment with bevacizumab combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years or older
* ECOG ≤2
* histologically proven unresectable metastatic colorectal adenocarcinoma
* Measurable lesion according to RECIST criteria
* Absence of prior chemotherapy for metastatic disease. Adjuvant chemotherapy following resection of the primary tumor is authorized if completed more than 6 months previously
* Patients treated with anticoagulants (coumadin, warfarin) can be included if close surveillance of the INR can be ensured. A change to low-molecular-weight heparin is preferable as long as the indications are respected
* Completed geriatric self-questionnaire
* Completed "Team" geriatric questionnaire (including Spitzer QoL Index)
* Written informed consent

Exclusion Criteria:

* Estimated life expectancy < 3 months
* Non-resolved intestinal occlusion or sub-occlusion
* Cerebral metastasis
* Other evolutive malignant tumor (non-stabilized cancer for less than 2 years)
* Evolutive gastroduodenal ulcer, wound or bone fracture
* Active heart disease: uncontrolled hypertension, myocardial infarction In the previous 6 months, angina, non-compensated congestive heart failure
* Major surgery, except for biopsy, or irradiation in the 4 weeks preceding the start of treatment
* Polynuclear neutrophils <1500/mm3, platelets <100 000/mm3 or 24-h proteinuria > 1g
* History of arterial thromboembolic event (cerebrovascular accident, transient ischemic attack, subarachnoid hemorrhage) in the 12 months preceding the first dose of bevacizumab
* History of distal or visceral ischemia ≥ grade 2 in the 12 months preceding the first dose of bevacizumab
* History of life-threatening pulmonary embolism in the 6 months preceding the first dose of bevacizumab
* Impossibility to ensure regular follow-up

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Initial examination | 21 days before the first course of treatment
  thoraco-abdomino-pelvic tomodensitometry or thoracic tomodensitometry and abdomino-pelvic MRI with identification and measurement of the target tumors according to RECIST (Response Evaluation Criteria in Solid Tumors
  )criteria.

SECONDARY OUTCOMES:
Initial examination | 14 days before inclusion
  Medical history, clinical examination (HR, arterial blood pressure
  , temperature, weight, height, Eastern Cooperative Oncology Group performance status),
  * measurement of body surface area, ECG
  * completion of questionnaire by the patient (annexe 1),
  * completion of geriatric questionnaire "team" (annexe 2)
  * biological examination including:
    * full blood count-platelets
    * blood electrolyte panel, creatinemia
    * Albumin
    * ASAT, ALAT, PAL, GGT, total and conjugated bilirubin
    * CEA, CA 19.9, LDH markers
    * balanced INR for patients on AVK
    * Urinary dip with 24-hour proteinuria if > 1+
  * Measurement of creatinine clearance using the Cockcroft formula (in men: (140-age) x weight (kg)/0.814 x creatinemia (μmol), in women: (140-age) x weight (kg)/0.85 x creatinemia (μmol)),
  * In the absence of a cardiological examination in the year before or in the case of a history of severe cardiovascular disease: consultation in cardiology.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Derived] Dohan A, Gallix B, Guiu B, Le Malicot K, Reinhold C, Soyer P, Bennouna J, Ghiringhelli F, Barbier E, Boige V, Taieb J, Bouche O, Francois E, Phelip JM, Borel C, Faroux R, Seitz JF, Jacquot S, Ben Abdelghani M, Khemissa-Akouz F, Genet D, Jouve JL, Rinaldi Y, Desseigne F, Texereau P, Suc E, Lepage C, Aparicio T, Hoeffel C; PRODIGE 9 Investigators and PRODIGE 20 Investigators. Early evaluation using a radiomic signature of unresectable hepatic metastases to predict outcome in patients with colorectal cancer treated with FOLFIRI and bevacizumab. Gut. 2020 Mar;69(3):531-539. doi: 10.1136/gutjnl-2018-316407. Epub 2019 May 17. PMID 31101691